CLINICAL TRIAL: NCT05916170
Title: Communicating Waterpipe Tobacco Harms to Reduce Use Among Young Adults: A Study of Hookah Café Customers in the Atlanta Area
Brief Title: A Study of Hookah Café Customers in the Atlanta Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB00095123; R01CA241420 (NIH)
Record Dates: First submitted 2023-05-10; First posted 2023-06-23 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2024-03

CONDITIONS: Waterpipe Tobacco Smoking
Keywords: Waterpipe Tobacco Smoking; Tobacco Smoking; waterpipe smoking behavior
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Intervention Model Description: The design of the study is a cluster randomized crossover trial, where the hookah café is the cluster and randomization is at the cluster level. Each hookah café will serve as its own control and will be used for data collection for both arms of the study. Cafes will start in the no-warning control arm and then will cross over to the intervention arm, where they will display one of four text-only warning signs. Participants will only participate in one of the arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Health Warnings (Experimental): Cafes will display text-only warning signs
  Interventions: Behavioral: Health Warnings
- Control - No Warnings (Experimental): No warnings posted in the hookah café
  Interventions: Behavioral: No Warnings

INTERVENTIONS:
Behavioral: Health Warnings — Text-only warnings about one health harm will be displayed in the hookah cafés where data collection is being conducted.
  Arms: Intervention - Health Warnings
Behavioral: No Warnings — No warnings posted in the hookah café
  Arms: Control - No Warnings

SUMMARY:
The purpose of the study is to assess the effectiveness of health warnings on waterpipe smoking behavior in a real-world setting. The primary hypothesis is that hookah café customers who are in the intervention (warning) arm will smoke less than customers who are in the control (no warning) arm, determined by differences in the boost in expired carbon monoxide from café entry to after café exit.

DETAILED DESCRIPTION:
Expired carbon monoxide is an objective biological marker of combustible tobacco smoking and is strongly correlated with the amount of smoke inhaled. In the intervention arm, warning messages will be displayed at various agreed-upon locations in the café, such as on hookah pipes, tables, countertops, walls, and menus. The goal is to maximize the potential for customers to be exposed to warnings. Participants will be patrons of the café and will be recruited before entering the café. Participants will complete a brief survey and provide a breath sample to measure expired carbon monoxide. When leaving the café, they will complete another survey and provide a second breath sample.

ELIGIBILITY:
Inclusion Criteria:

* Planning to enter the hookah café where study is being conducted
* Age 18 or older
* English speaking
* Planning to smoke hookah inside
* Not planning to smoke cigarettes, cigars, cigarillos or marijuana while at the hookah café
* Had not previously entered the café earlier in the day on the same day/night as data collection
* Has not been approached to participate in the study at another café or another day/night at the current café
* Are not employees of the business
* Have capacity to participate as determined by the staff member conducting eligibility screening

Exclusion Criteria:

* Not planning to enter the hookah café where the study is being conducted
* Age 17 and under
* Non-English speaking
* Not planning to smoke hookah in the café
* Planning to smoke cigarettes, cigars, or marijuana while at the hookah café
* Are employees of the business
* Had previously entered the café on the same day/night as data collection
* Has not been approached to participate in the study previously
* Does not have capacity to participate as determined by the staff member conducting eligibility screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 977 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-21 (Actual); Study Completion 2024-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Sutfin, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a cluster randomized crossover trial in which hookah cafes started in the No Warning Control condition and then crossed over to the Health Warnings Intervention, in which they were randomized to display one of four health warning messages (Milestones). Participants were cafe patrons on the days/nights that data collection was being conducted. Participants were only permitted to participate in one instance of data collection at one hookah cafe. Some cafes only had Control period.
Pre-assignment Details: The Control and Intervention arms are reported as two periods in a single arm for this crossover study. The total enrollment to the study across both periods was 977. 507 participants were enrolled during the Control period of the cafes and 470 were enrolled during the Intervention period. Participants did not participate in more than one period.
Units Other Than Participants: Hookah Cafe
Groups:
- Hookah Cafes in Atlanta, GA: Each hookah café will serve as its own control and will be used for data collection for both arms of the study. Cafes will start in the no-warning control arm and then will cross over to the intervention arm, where they will display one of four text-only warning signs. Participants will only participate in one of the arms.
Period: No Warning Control
Arm/Group | Hookah Cafes in Atlanta, GA
Started | 507; 27 Hookah Cafe
Completed | 479; 27 Hookah Cafe
Not Completed | 28; 0 Hookah Cafe
Not completed — Lost to Follow-up | 12
Not completed — Withdrawal by Subject | 15
Not completed — Noncompliance with protocol | 1
Period: Health Warning Intervention
Arm/Group | Hookah Cafes in Atlanta, GA
Started | 470; 23 Hookah Cafe
Lung Damage Warning | 148; 6 Hookah Cafe
Heart Damage Warning | 104; 5 Hookah Cafe
CO Poison Warning | 112; 6 Hookah Cafe
Fetal Damage Warning | 106; 6 Hookah Cafe
Completed | 431; 19 Hookah Cafe
Not Completed | 39; 4 Hookah Cafe
Not completed — Lost to Follow-up | 15
Not completed — Withdrawal by Subject | 10
Not completed — Noncompliance with protocol | 14

BASELINE CHARACTERISTICS:
Groups:
- No Warning Control: No warnings posted in the hookah café
  No Warnings: No warnings posted in the hookah café
- Health Warning Intervention: Cafes will display text-only warning signs
  Health Warnings: Text-only warnings about one health harm will be displayed in the hookah cafés where data collection is being conducted.
- Total: Total of all reporting groups
Arm/Group | No Warning Control | Health Warning Intervention | Total
Number analyzed (Participants) | 507 | 470 | 977
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.9 (6.9) | 31.5 (7.3) | 31.2 (7.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 295 | 289 | 584
  Male | 203 | 177 | 380
  Unknown | 9 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 26 | 61
  Not Hispanic or Latino | 458 | 427 | 885
  Unknown or Not Reported | 14 | 17 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 6 | 10
  Asian | 38 | 28 | 66
  Native Hawaiian or Other Pacific Islander | 4 | 0 | 4
  Black or African American | 389 | 380 | 769
  White | 12 | 14 | 26
  More than one race | 23 | 19 | 42
  Unknown or Not Reported | 37 | 23 | 60
Region of Enrollment [Number; unit: participants]
  United States | 507 | 470 | 977

OUTCOME MEASURES:

1. Primary Outcome: Change in Expired Carbon Monoxide (eCO Boost)
Description: Change in eCO from baseline (before entry into the hookah café) to follow-up (upon exit from the hookah café) - eCO will be measured with the Bedfont Micro+ Smokerlyzer. Higher scores represent higher concentrations of Carbon Monoxide (CO), which is correlated with greater waterpipe use.
Time Frame: Baseline and after exiting the café up to 10 hours
Population: Participants were included in analysis if they completed both pre- and post-cafe eCO collection in cafes that completed both the control and intervention arms of this crossover trial. Participants in each arm are unique.
Measure: Mean (Standard Error); unit: parts per million
Groups:
- No Warning Control: No warnings posted in the hookah café
- Health Warning Intervention: Each cafe displayed signs communicating one of four health warning messages. The primary outcome is reported as all of the health warnings aggregated versus the no warning control.
Arm/Group | No Warning Control | Health Warning Intervention
Number analyzed (Participants) | 356 | 375
parts per million | 25.7 (2.93) | 23.5 (2.91)

2. Other Pre Specified Outcome: Behavioral Intention
Description: Participants will be asked at three items assessing their anticipated hookah smoking within the next month. Items will be averaged to create a composite score of intent to continue the behavior within the next month.
  1. How interested are you in smoking tobacco in a hookah in the next month?
  2. How likely are you to smoke tobacco in a hookah in the next month?
  3. How much do you plan to smoke tobacco in a hookah in the next month? Response options: (1) Not at all, (2) Very little, (3) Somewhat, (4) Quite a bit, (5) Very much
Time Frame: at exit; up to 10 hours
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Quit Motivation
Description: One item to measure participants' motivation to quit smoking hookah, rated on a 1-10 scale of Not at all motivated to Extremely motivated
Time Frame: at exit; up to 10 hours
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Hookah Use Behavior
Description: Participants will be asked a variety of items to assess their hookah smoking behaviors within the café. Items will be scored individually.
  1. Did you smoke hookah in this café/lounge/bar today? (1) Yes, (2) No
  2. (If no) Why didn't you smoke hookah in this café/lounge/bar today? Free text response
  3. (If yes) Compared to a typical night, how much did you smoke? (1) Less hookah than usual, (2) About the same amount of hookah as usual, (3) More hookah than usual, (4) This was my first time smoking hookah
  4. (If less) Why did you smoke less than usual? Free text response
  5. (If more) Why did you smoke more than usual? Free text response
Time Frame: at exit; up to 10 hours
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Subjective Experiences of Smoking Hookah
Description: Eight items from the Product Evaluation Scale (Hatsukami et al. 2013) will be used to assess participants' subjective experiences of smoking hookah. Items scores will be averaged across the subscale.
  1. Was it satisfying?
  2. Did it taste good?
  3. Did you enjoy the sensations in your mouth?
  4. Did you enjoy it?
  5. Did it make you dizzy?
  6. Did it make you nauseous?
  7. Was it too much nicotine?
  8. Were there bothersome side effects? Response options: (1) Not at all - (7) Extremely
Time Frame: at exit; up to 10 hours
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Knowledge
Description: Four items to assess participants' knowledge of health harms based on warning statements used across the study. We will calculate a sum score for each individual with higher scores indicating more accurate knowledge.
  Response options: True / False / I don't know
Time Frame: at exit; up to 10 hours
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Beliefs
Description: Four items to assess the participants' agreement with statements of how each of the four health harms utilized across the study apply to their own health. We will calculate a mean score across all four items for each individual, where higher scores indicate stronger beliefs about personal harm from hookah smoking.
  Response options: (1) Strongly disagree to (5) Strongly agree
Time Frame: at exit; up to 10 hours
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Warning Recall
Description: One Y/N item to assess participants' exposure to warnings. If participants report warning exposure, an open-ended item will assess warning recall.
Time Frame: at exit; up to 10 hours
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Warning Recognition
Description: Participants in the intervention arm will be asked to select the warning(s) that they saw at the café from four possible warnings. For each warning message that they report having seen, they will be asked to select where they saw the warning from a list of possible locations. (Intervention arm only)
Time Frame: at exit; up to 10 hours
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Social Interaction
Description: For each warning selected in the Warning Recognition section, participants will be asked if they discussed the warning with others. If they answer positively, they will be given a list of topics to choose from to describe what they talked about, including a free-text option.
Time Frame: at exit; up to 10 hours
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Perceived Influence of Warning on Smoking Behavior Answers
Description: Participants will be asked whether they changed their smoking behavior as a result of the warning(s) they saw (as reported in the Warning Recognition section). They will be asked to report whether they smoked more, less, or the same amount as they usually do. These items will be asked for each warning the participant reports seeing.
Time Frame: at exit; up to 10 hours
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Time Spent in the café
Description: Duration of time in café will be calculated from the time of completion of eCO measurement at Time 1 to start of survey at Time 2. Additionally, we will utilize a subjective measure of time spent in the café: Compared to what you planned, how long did you stay at the café/lounge/bar? (Longer, shorter, about the same).
Time Frame: at exit; up to 10 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the time that the participant was in the cafe, approximately 3 hours.
Arm/Group | Control - No Warnings | Intervention - Health Warnings
All-Cause Mortality (participants affected / at risk) | 0/507 | 0/470
Serious Adverse Events (participants affected / at risk) | 0/507 | 0/470
Other Adverse Events (participants affected / at risk) | 0/507 | 0/470

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT05916170/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT05916170/ICF_000.pdf